CLINICAL TRIAL: NCT06628011
Title: Digital Follow-up of Exercise Training in Outpatients With Mental Disorders
Brief Title: Digital Follow-up of Aerobic Interval Training in Outpatients With Mental Disorders
Acronym: DIG-EX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Molde University College (Other); NTNU Health (sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 633068
Record Dates: First submitted 2024-08-15; First posted 2024-10-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Severe Mental Disorder
Keywords: Peak oxygen uptake; Aerobic high-intensity interval training; Digital follow-up; Mental health disorder; Exercise physiology
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a 1:1 allocation ratio into an Intervention Group or Control Group.
Masking Description: Participants are aware of which group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will be encouraged to perform two aerobic interval training sessions per week for 12 weeks, on their own and not at the exercise training clinic, while receiving digital follow-up support through HelsaMi and exercise guidance through the exercise app. The digital follow-up through HelsaMi will consist of overview of treatment progress and schedule, communication with health care personnel (video consultation or chat up to 2 times per week), notifications reminding them to exercise, exercise diary, questionnaires, and educational content.
  Interventions: Other: Intervention group/training group
- Control gorup (No Intervention): This group will be encouraged to perform the same exercise training but without any follow-up support

INTERVENTIONS:
Other: Intervention group/training group — We will assess the short-term effects through a 12-week intervention, and its long-term effects after 1-year. Both the intervention group (IG) and control group (CG) will receive two sessions of aerobic interval training at the Exercise Training Clinic, situated at the Department of Psychosis and Rehabilitation, Psychiatry Clinic, St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway. One training session consists of 36 minutes of high intensity training (HIT).
  Arms: Intervention group

SUMMARY:
This randomized-controlled trial (RCT) will investigate if digital follow-up of exercise, i.e. followup through the new citizen portal HelsaMi, coupled with an exercise app can result in exercise adherence and improved oxygen uptake in individuals with mental disorders (MD). Secondary, the project will provide information regarding effects on cardiovascular disease risk-factors, functional capacity, quality of life, satisfaction, and cost through a randomized-controlled trial (RCT) including individuals with MDs.

Outcomes assessed in this project, such as maximal oxygen uptake, functional capacity, and quality of life, are strongly related to the ability to carry out activities of daily living. These outcomes are associated with benefits such as reduced sick leave, extended life expectancy, independence, and improved health status with increasing age. Economically, with the world population growing older and health care resources being stretched, there is clearly a need to apply and evaluate effective alternative methods to improve somatic health on a broader scale in a sustainable fashion, preferably utilizing existing platforms and exercise apps.

DETAILED DESCRIPTION:
The main aim of this randomized controlled trial (RCT) is to investigate if digital exercise followup can support exercise adherence and result in increased aerobic capacity in individuals with MDs. We will assess the short-term effects through a 12-week intervention, and its long-term effects after 1-year. Both the intervention group (IG) and control group (CG) will receive two sessions of aerobic interval training at the Exercise Training Clinic, situated at the Department of Psychosis and Rehabilitation, Psychiatry Clinic, St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway. One training session consists of 36 minutes of high intensity training (HIT). HIT consists of 4x4 intervals on a treadmill at 85-95% of maximal heart rate, interspersed by 3minute active rest periods at 70% maximal heart rate [31]. Following the educational exercise sessions at the Exercise Training Clinic, the IG will be encouraged to perform two aerobic interval training sessions per week for 12 weeks, on their own and not at the exercise training clinic, while receiving digital follow-up support through HelsaMi and exercise guidance through the exercise app. The digital follow-up through HelsaMi will consist of overview of treatment progress and schedule, communication with health care personnel (video consultation or chat up to 2 times per week), notifications reminding them to exercise, exercise diary, questionnaires, and educational content.

Objective. To investigate if digital exercise follow-up through HelsaMi combined with an exercise app (Myworkout GO) in individuals with MDs is more effective at improving exercise adherence and aerobic capacity compared to standard treatment coupled with advice on how to perform high intensity interval training without any digital follow-up.

Main hypothesis. Digital follow-up of exercise yields better results than only being advised to exercise at improving exercise adherence, peak oxygen uptake (V̇ O2peak), work efficiency, functional capacity, and quality of life after 12 weeks and 1-year.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving outpatient mental health treatment at the clinics of mental health at St. Olavs Hospital,.

  .-18-65 years old
* Both men and women able to carry out exercise training.
* Participants must be capable of giving informed consent and use HelsaMi.

Exclusion Criteria:

* Contraindications for exercise training and testing according to the ACSM specifications; life-threatening or terminal medical conditions; unable to carry out intervention or test procedures; pregnancy; mothers <6 months post-partum.
* Inpatients at an acute psychiatric ward or have any planned surgery that would interfere with the intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | Baseline, 12 weeks, 1 year
  Peak oxygen uptake after the training period subtracted Peak oxygen uptake at baseline. Using the The Vyntus ONE with a mixing chamber. It is a powerful tool for comprehensive cardiopulmonary testing, providing accurate and reliable data to help clinicians make informed decisions.

SECONDARY OUTCOMES:
Physical activity measurement | 1-2 weeks
  Physical activity level for 1-2 weeks (triaxial accelerometer, wGT3X-BT, ActiGraph LLC, USA)
Use of health care services | Baseline, 12 weeks, 1 year
  Medical record data, Norwegian patient register (NPR) and the Norwegian Registry for Primary Health Care (NRPHC) - which together cover all governmental-funded health care, and occupational status (NAV)
Usage data of HelsaMi | Baseline, 12 weeks, 1 year
  Helseplattformen: Number of times logging in, time spent in the program. Usaga data from the exercise app such as number of exercise sessions logged, and exercise intensity will be collected from Myworkout AS. Medications, diagnosis, number of hospitalizations
Functional performance/capacity | Baseline, 12 weeks, 1 year
  * Sit-to-stand test: 30-second sit-to-stand test. Number of full stands in 30 seconds.
  * Unipedal stance test: Single leg stance. Measured in seconds.
  * Stair performance: Stair test. Participants are instructed to ascend and descend 18 steps 3 consecutive times. Performance measured in seconds.
Feasibility - Drop-out/retention | 12 weeks, 1 year
  Follow-up through HelsaMI. Training session diary of exercise performed from the Myworkout GO app.
Changes in walking economy | Baseline, 12 weeks, 1 year
  Walking economy (oxygen uptake at a standard workload) after the training period subtracted walking economy at baseline. It is tested at a submaximal workload and calculated as a reduction in whole body pulmonary V̇O2 or energy expenditure (Kcal∙-min) accomplished during walking.
Motivation to Exercise: Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) | Baseline, 12 weeks, 1 year
  The BREQ-2 is a 19-item questionnaire that measures different types of motivation for exercise based on self-determination theory. It includes factors such as intrinsic motivation, identified regulation, introjected regulation, external regulation, and amotivation
Health Literacy: eHealth Literacy Scale (eHEALS) | Baseline, 12 weeks, 1 year
  The eHEALS is an 8-item scale designed to assess consumers' perceived skills at finding, evaluating, and applying electronic health information. It measures knowledge, comfort, and perceived skills in using eHealth resources
Mental Health-Related Barriers and Benefits to Exercise: MEX | Baseline, 12 weeks, 1 year
  The MEX scale is a 30-item measure that assesses mental health-related barriers and benefits to exercise. It includes two subscales: one for barriers and one for benefits, each with 15 items. It is designed to understand how mental health symptoms impact exercise engagement.
Potential Barriers and Enablers Reported: System Usability Scale (SUS) | Baseline, 12 weeks, 1 year
  The SUS is a 10-item Likert scale that provides a global measure of system usability. It assesses the effectiveness, efficiency, and satisfaction of a system from the user's perspective
Patient satisfaction (questionnaires) | Baseline, 12 weeks, 1 year
  Client Satisfaction Questionnaire-8 (CSQ-8): The CSQ-8 is an 8-item questionnaire designed to measure client satisfaction with health and human services. It provides a global measure of satisfaction, with items rated on a 4-point scale from "1" (low satisfaction) to "4" (high satisfaction).
Patient activation | Baseline, 12 weeks, 1 year
  Patient Activation Measure for Mental Health (PAM-13, MH): The PAM-13 is a 13-item questionnaire that assesses a patient's knowledge, skills, and confidence in managing their own health. It is specifically adapted for mental health contexts to measure the level of patient activation
Quality of life | Baseline, 12 weeks, 1 year
  Quality of life: SF-36® Health Survey (SF-36): Designed to measure overall health status and quality of life. It covers eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health
Quality-adjusted life year | Baseline, 12 weeks, 1 year
  EuroQol five dimensions questionnaire (EQ-5D-3L): A standardized instrument used to measure health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with three levels of severity. It also includes a visual analogue scale (VAS) for self-rated health.

OTHER OUTCOMES:
Body composition | Baseline, 12 weeks, 1 year
  Body weight, measured in kilograms (kg). Height, measure in centimeters (cm). Body mass index (BMI) calculated by dividing the weight in kilograms by the square of the height in meters. Waist Circumference, Waist circumference is the measurement taken around the abdomen at the level of the belly button. It is used to assess abdominal fat.
Blood pressure | Baseline, 12 weeks, 1 year
  The force of blood pushing against the walls of the arteries. It is measured using two numbers: systolic pressure (when the heart beats) and diastolic pressure (when the heart rests between beats).
Blood Samples | Baseline, 12 weeks, 1 year
  Glucose: Measures the level of sugar in the blood. It is used to diagnose and monitor diabetes. Triglycerides: Measures the amount of fat in the blood. High levels can increase the risk of heart disease. HbA1C: Measures the average blood sugar levels over the past 2-3 months. It is used to diagnose and monitor diabetes. Apolipoprotein A1: The main protein component of HDL (good cholesterol). It helps in the transport of cholesterol from tissues to the liver.
  Apolipoprotein B: The main protein component of LDL (bad cholesterol). It is involved in the transport of cholesterol to tissues and is a marker for cardiovascular risk. Cholesterol: High-Density Lipoprotein (HDL): Known as "good" cholesterol, it helps remove bad cholesterol from the bloodstream.
  Low-Density Lipoprotein (LDL): Known as "bad" cholesterol, high levels can lead to plaque buildup in arteries and increase the risk of heart disease. Total Cholesterol: The sum of HDL, LDL, and other lipid components in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- St. Olavs Hospital HF. And NTNU (Norwegian University of Science and Technology) Department of Mental Health, Faculty of Medicine and Health Sciences, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No